CLINICAL TRIAL: NCT02516878
Title: Acupuncture for Body Weight Control: A Pilot Randomized Controlled Trial
Brief Title: Acupuncture for Body Weight Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, ZhaoXiang Bian, Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AcupBWC001
Record Dates: First submitted 2015-07-30; First posted 2015-08-06 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: acupuncture; Chinese Medicine; obesity
MeSH Terms: conditions — Obesity | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture group (Experimental): Eight body acupuncture points will be chosen as Tianshu(ST-25), Daheng(SP-15), Daimai(GB-26), Qihai(CV-6), Zhongwan(CV-12), Zusanli(ST-36), Fenlong(ST-40), Sanyinjiao(SP-6). The needles will be retained for 30 minutes.
  Participants of the treatment group will additionally receive unilateral auricular acupressure at four auricular points as Hunger, Shen men, Spleen and Stomach with Semen Vaccariae embedded within adhesive tape in each treatment session. Acupressure will be applied by the subjects with repeat pressing of the tape with fingertips for 3 minutes per point, 3 times per day. The embedded tape will be retained in-situ until the next visit and then the alternate side of ear will be treated.
  Interventions: Procedure: Acupuncture
- Control group (Sham Comparator): For subjects assigned to control group, Streitberger's non-invasive acupuncture needles (Gauge 8 x 1.2" / 0.30 x 30 mm) will be applied to serve as sham control at the same acupoints with the same stimulation modality, except that the needles are only adhered to the skin instead of insertion.
  The Semen Vaccariae embedded tape used in treatment group will be applied on 4 non-acupoints at the helix unilaterally, retained until the next visit and then the alternate ear will be used.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Eight body acupuncture points will be chosen as Tianshu(ST-25), Daheng(SP-15), Daimai(GB-26), Qihai(CV-6), Zhongwan(CV-12), Zusanli(ST-36), Fenlong(ST-40), Sanyinjiao(SP-6). The needles will be retained for 30 minutes.
  Participants of the treatment group will additionally receive unilateral auricular acupressure at four auricular points as Hunger, Shen men, Spleen and Stomach with Semen Vaccariae embedded within adhesive tape in each treatment session. Acupressure will be applied by the subjects with repeat pressing of the tape with fingertips for 3 minutes per point, 3 times per day. The embedded tape will be retained in-situ until the next visit and then the alternate side of ear will be treated.

SUMMARY:
In this study, a 18-week, single-blinded, randomized controlled clinical trial will be conducted to evaluate the effectiveness, efficacy and safety of acupuncture on weight control in Hong Kong.

DETAILED DESCRIPTION:
This is a pilot single-blind, randomized, sham-controlled trial. 72 participants will be randomly assigned to acupuncture group or control group. The duration of the treatment will be 8 weeks with 2 sessions per week and the follow-up period will be 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65 years old;
* body mass index (BMI)≥25 kg/m2;
* having not received any other weight control measures or any medical and/or drug history within the last 3 months.

Exclusion Criteria:

* endocrine diseases;
* heart diseases;
* patients with pacemaker;
* allergy and immunology diseases;
* having bleeding tendency;
* pregnant or lactating women;
* having impaired hepatic or renal function;
* stroke or otherwise unable to exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in body weight during treatment and follow up | The change in body weight will be assessed every two weeks during 8-week treatment and 8-week follow up
  measured by Omron KARADA Scan Body Composition & Scale

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) during treatment and follow up | The change in BMI will be assessed every two weeks during 8-week treatment and 8-week follow up
  The change in Body Mass Index (BMI) will be measured by Omron KARADA Scan Body Composition & Scale
Change in waist circumference during treatment and follow up | The change in waist circumference will be assessed every two weeks during 8-week treatment and 8-week follow up
Change in hip circumference | The change in hip circumference will be assessed every two weeks during 8-week treatment and 8-week follow up
Change in body fat percentage during treatment and follow up | The change in body fat percentage will be assessed every two weeks during 8-week treatment and 8-week follow up
  The change in body fat percentage will be measured by Omron KARADA Scan Body Composition & Scale
Number of patients with adverse events after treatment | Number of patients with adverse events after treatment will be recorded and compared among the two groups during 8-week treatment and 8-week follow up

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoxiang Bian, MD., Ph.D, Study Director — Hong Kong Baptist University

REFERENCES:
- [Derived] Zhong LL, Kun W, Lam TF, Zhang SP, Yang JJ, Ziea TC, Ng B, Bian ZX. The combination effects of body acupuncture and auricular acupressure compared to sham acupuncture for body weight control: study protocol for a randomized controlled trial. Trials. 2016 Jul 25;17(1):346. doi: 10.1186/s13063-016-1458-2. PMID 27457720